CLINICAL TRIAL: NCT05696860
Title: The Effect of Microstream® Capnography on Patient Safety in Endobronchial Ultrasonography Applications Under Sedation
Brief Title: Microstream® Capnography in Endobronchial Ultrasonography Applications Under Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Sinem Cetinkaya Ozpar, Doctor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BUU2019/8-18
Record Dates: First submitted 2022-12-26; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Capnography; Endobronchial Ultrasound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitorization with Capnography (Experimental): Patients followed with capnography and standard monitorization
  Interventions: Device: Capnography Monitoring
- Monitorization Without Capnography (No Intervention): Patients followed with standard monitorization

INTERVENTIONS:
Device: Capnography Monitoring — Capnography monitoring
  Arms: Monitorization with Capnography

SUMMARY:
Purpose: Researchers wanted to investigate the effect of capnography monitoring in addition to routine monitoring on the development of desaturation and other vital parameters in endobronchial ultrasonography (EBUS) cases.

Method: 100 patients who underwent EBUS under sedation will be included in this prospective and randomized controlled study. The cases will be divided into two groups of 50 people each. In the first group, standard monitoring will be performed, and in the second group, in addition to standard monitoring, capnography monitoring will be used. Heart rate, blood pressure, peripheral oxygen saturation (SpO2) values in both groups, end-tidal carbon dioxide (EtCO2), respiratory rate and integrated pulmonary index (IPI) values in the second group will be recorded in all cases. Disturbances in vital parameters and airway interventions, which were common in both groups, will ve compared. The frequency of problems detected by capnography monitoring in the second group will be examined.

DETAILED DESCRIPTION:
Endobronchial ultrasonography (EBUS) is an examination method that has been increasingly used in diagnosing and staging lung cancer, mediastinal lymphadenopathy and masses in recent years. This procedure is performed under anesthesia. General anesthesia or sedation is generally preferred as an anesthesia option. Desaturation may frequently develop during this procedure. Follow-up with standard perioperative monitoring methods (heart rate - HR, respiratory rate - SS, peripheral oxygen saturation - SpO2) is not a proper approach to detecting respiratory depression before desaturation develops.

Capnography is a monitoring method that detects respiratory depression before desaturation develops by making instant end-tidal carbon dioxide (EtCO2) measurements. It has been stated that it significantly reduces the risk of desaturation in many surgical and interventional procedures performed under sedation and general anesthesia. In addition, respiratory disorders such as bronchospasm, apnea or hypopnea can be detected by capnography. However, there is no information about capnography's effect on desaturation development or its contribution to standard monitoring in EBUS cases.

The purpose of this study was to investigate the effects of capnography monitoring in addition to routine monitoring on the development of desaturation and other vital parameters in EBUS cases under moderate sedation according to the Ramsay Sedation Scale (RSS). The primary aim was to compare the groups in terms of the development of desaturation, and the secondary aim was in terms of duration of hypoxemia, development of severe hypoxemia, lowest SpO2 value, development of hypotension, and bradycardia.

150 patients who will undergo elective EBUS procedure, have scores between 1-3 according to the American Society of Anesthesiologists (ASA) classification, are pregnant or not suspected of pregnancy, approve the informed consent form, and are not allergic to the sedation agents to be used, will be included in the study. Patients with an ASA score of 4 and above, pregnant or suspected pregnancy, patients with difficult airway features, and emergency cases will be excluded from the study.

The cases will be divided into two groups of 75 people using the closed envelope method. There will be cases in which capnography monitorization was performed in group 1 (experimental group), and cases in which capnography monitoring was not performed in group 2 (control group). In all cases, age, gender, weight, height, ASA class, doses of applied anesthesia drugs, and smoking history will be recorded. After obtaining informed consent in all cases Standard monitoring and BIS monitoring will be performed before sedation, including HR, SS, SpO2, BP, and 3-lead electrocardiographic analysis. In addition to standard monitoring in patients in Group 1, ETCO2, integrated pulmonary index (IPI) will be measured non-invasively prior to sedation through a nasal cannula (FilterLine®) connected to the capnography device (Capnostream® 20p). Sedation and analgesia will be performed in accordance with the routine sedation-analgesia protocol used by our department in EBUS cases. There will be no changes to the routine protocol. In accordance with this protocol, after the patient is taken to the operating room, 5 ml of 2% lidocaine will be applied with a reservoir mask for topical anesthesia. As a sedative agent, 1-2 mg of midazolam will be administered intravenously. A nasopharyngeal airway will be placed and 5 lt/min oxygen will be given to all patients throughout the operation. In induction, remifentanil will be administered at a level of 0.04 µg/kg/min and Propofol at a level of 0.5-1 mg/kg/hour. The target sedation level will be determined as 60-80 BIS score and will be level 3 (moderate sedation, sleepy but responsive to verbal stimuli) according to the Ramsey Sedation Scale. All parameters measured before sedation in both groups; It will be recorded at 3 minutes, 6 minutes, 9 minutes after sedation, and at 3-minute intervals until the end of the operation.

During the operation, in the cases in Group 1, apnea (the ETCO2 waveform is not seen for 10 seconds), hypopnea (at least 50% decrease in the peak ETCO2 level in 2 consecutive waveforms compared to the initial value and the peak ETCO2 level in the second wave is lower than the first) and the number of bronchospasm, The number of episodes of cough, tachycardia, bradycardia, hypoxemia (SpO2<90%) in both groups, duration of anesthesia, duration of the procedure (time between insertion and removal of the bronchoscope) and recovery time (spontaneous opening of the eyes of the patients with the removal of the bronchoscope, performing the finger-nose test) and the time elapsed between the time he was able to tell his birth dates) will be recorded. If bronchospasm, upper airway obstruction, apnea, bradypnea develop during the procedure, jaw-thrust maneuvers, head-tilt maneuvers, verbal and tactile warnings will be recorded.

After the operation, the cases will be taken to the recovery unit. From the moment of entry in the recovery unit; BP, EtCO2, SpO2 and IPI values will be recorded every 5 minutes until the exit time. In accordance with the routine sobering protocol; Patients with a Modified Aldrete Score of 9 or higher will be sent to the clinic.

The frequency and interrelationship of the parameters evaluated in both groups will be examined. Between the group that underwent capnography and the group that did not; It will be investigated whether there is a significant difference in terms of apnea, desaturation episodes and interventions.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score of 1-3,
* No pregnancy or suspected pregnancy
* No allergy history
* Signed informed consent

Exclusion Criteria:

* Emergency EBUS cases
* ASA score of 4
* Allergy or pregnancy history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Desaturation Development - Peripheric oxygen saturation decrease less than 90% on Pulse Oximetry | During Sedation, an average of 1 hour
  Compare Experimental and Control Groups in Terms of Desaturation Development

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Nur Kaya, Study Director — Supervisor
Locations (1):
- Bursa Uludag University Department of Anesthesiology and Reanimation, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No